CLINICAL TRIAL: NCT07150286
Title: Assessment of Hematological Effect of H.Pylori and H.Pylori Eradication Therapy Among a Sample of Iraqi ITP Patients
Brief Title: Helicobacter Pylori Eradication Therapy for Immune Thrombocytopenia (ITP) Patients in Iraq
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Mustansiriyah University (Other)
Responsible Party: Principal Investigator, Murtadha Al-Owayef, Murtadha Salah Shyaa Al-OWAYEF, Al-Mustansiriyah University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 96
Record Dates: First submitted 2025-08-24; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Immune Thrombocytopenic Purpura; HELICOBACTER PYLORI INFECTIONS
Keywords: immune thrombocytopenia; ITP; Helicobacter pylori; H.pylori; Levofloxacin-based Triple Therapy; Salvage Therapy; Hematology; Iraq
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Intervention Model Description: This is a two-arm, parallel-group study. Patients with ITP who test positive for H. pylori receive a 14-day levofloxacin-based eradication regimen, while H. pylori-negative ITP patients serve as the comparison group without eradication therapy. Platelet counts are monitored before and after treatment to assess hematological response.
Masking Description: This is an open-label study. All participants, investigators, and care providers are aware of group assignments, as treatment allocation is based on H. pylori infection status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- H. pylori-Positive ITP Patients - Eradication Therapy (Experimental): Patients who test positive for Helicobacter pylori will receive a 14-day levofloxacin-based triple therapy regimen according to ACG guidelines. Platelet counts will be measured at baseline and four weeks after completion of therapy to assess hematological response.
  Interventions: Drug: Levofloxacin-Based H. pylori Eradication Therapy
- H. pylori-Negative ITP Patients - No Therapy (No Intervention): Patients who test negative for H. pylori will not receive eradication therapy. Platelet counts will be monitored at the same time points as the intervention group to serve as a comparison for evaluating treatment effects.

INTERVENTIONS:
Drug: Levofloxacin-Based H. pylori Eradication Therapy — This intervention consists of a 14-day levofloxacin-based triple therapy regimen for Helicobacter pylori eradication in ITP patients. The regimen follows current ACG guidelines and typically includes:
  Levofloxacin - antibiotic targeting H. pylori
  Amoxicillin - antibiotic used in combination for enhanced efficacy
  Proton Pump Inhibitor (PPI) - to reduce stomach acid and improve antibiotic effectiveness
  Patients will receive the full 14-day course, and platelet counts will be measured at baseline and four weeks post-therapy to assess hematological response. This intervention is unique to H. pylori-positive ITP patients in this study and is not administered to H. pylori-negative patients.
  Arms: H. pylori-Positive ITP Patients - Eradication Therapy

SUMMARY:
This study is being conducted to evaluate the effect of treating Helicobacter pylori infection on platelet counts in patients with immune thrombocytopenia (ITP). ITP is a condition in which the body's immune system attacks its own platelets, leading to an increased risk of bleeding and bruising. Some studies have suggested that removing H. pylori infection may help improve platelet counts in certain patients with ITP.

In this study, 100 patients with ITP will be enrolled at hematology centers in Baghdad. Patients will be tested for H. pylori infection using stool antigen testing. Those who are positive will receive a 14-day antibiotic treatment (levofloxacin-based therapy) to eradicate the infection. Platelet counts will be measured before and after therapy to determine whether successful eradication improves platelet levels.

The findings from this study may help provide new treatment options for ITP patients and give doctors in Iraq more evidence about how H. pylori infection affects blood disorders.

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP) is an acquired autoimmune disorder characterized by low platelet counts and increased bleeding risk. Several studies have suggested a link between Helicobacter pylori infection and platelet recovery following eradication therapy, though results differ across regions and populations.

This investigator-initiated, prospective study aims to assess the hematological effect of H. pylori eradication in Iraqi patients with ITP. A total of 100 patients will be recruited at two hematology centers in Baghdad. Patients will undergo stool antigen testing to determine H. pylori status.

The study is divided into two phases:

Phase 1: Observational cross-sectional analysis of ITP patients who are H. pylori negative.

Phase 2: Interventional, prospective, open-label evaluation of ITP patients who are H. pylori positive compared with H. pylori negative controls.

Patients testing positive for H. pylori will receive a 14-day levofloxacin-based triple therapy regimen consistent with current American College of Gastroenterology (ACG) guidelines. Platelet counts will be measured at baseline and four weeks after therapy completion. Outcomes will focus on hematological response to eradication, with secondary analysis comparing platelet recovery between H. pylori positive and negative patients.

This study is the first in Iraq to evaluate the impact of salvage therapy for H. pylori eradication in ITP patients. The results may provide novel insights into regional differences in treatment response and inform future clinical practice guidelines for managing ITP.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) with a confirmed diagnosis of ITP Platelet count <100,000/µL. H. pylori-positive or H. pylori-negative based on stool antigen test

Exclusion Criteria:

* • Patients with other causes of thrombocytopenia (e.g., leukemia, aplastic anemia).

  * Severe comorbidities (e.g., uncontrolled diabetes, severe cardiac disease).
  * Recent use (within 4 weeks) of antibiotics, proton pump inhibitors, or bismuth compounds.
  * Concurrent use of medications that interfere with H. pylori therapy or platelet levels.
  * Pregnant or lactating women.
  * Known allergy or intolerance to eradication therapy agents (clarithromycin, amoxicillin, metronidazole).
  * High risk of poor compliance (e.g., psychiatric illness).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Change in Platelet Count After H. pylori Eradication | Baseline and 4 weeks post-therapy
  The primary outcome is the absolute change in platelet count (×10⁹/L) from baseline to four weeks after completion of levofloxacin-based H. pylori eradication therapy in H. pylori-positive ITP patients. Platelet counts will be measured using standard hematology analyzers (Hemmary 86 and Cellagon 5 Pro).

CONTACTS AND LOCATIONS:
Overall Officials: Manal Khalid Abdulridha, proffessor at Mustansiriyah, Principal Investigator — Al-Mustansiriyah University - National Center of Hematology
Locations (1):
- Al-Mustansiriyah University - college of pharmacy - clinical pharmacy department, Baghdad, Baghdad Governorate, Iraq

IPD SHARING:
Plan to Share IPD: Undecided